CLINICAL TRIAL: NCT00164112
Title: Comparison of the Effect of Azithromycin, Telithromycin and Levofloxacin on Drug Metabolizing Enzymes Using the Validated Cooperstown 5+1 Cocktail
Brief Title: Comparative Effects of Azithromycin, Telithromycin and Levofloxacin on Drug Metabolizing Enzymes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CAPSS-273
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-03

CONDITIONS: Healthy
Keywords: Cooperstown Cocktail; Drug Metabolizing Enzymes; Drug Interactions; Phenotyping
MeSH Terms: interventions — Azithromycin; telithromycin; Levofloxacin

INTERVENTIONS:
Drug: Cooperstown 5+1 alone
Drug: Azithromycin plus Cooperstown 5+1
Drug: Telithromycin plus Cooperstown 5+1
Drug: Levofloxacin plus Cooperstown 5+1

SUMMARY:
Studies have previously shown that a broad drug interaction screening can be performed using enzyme specific probes such as oral caffeine for CYP1A2, N-acetyltrasferase-2 (NAT-2), and xanthine oxidase (XO), warfarin plus vitamin K for CYP2C9, omeprazole for CYP 2C19, dextromethorphan for CYP2D6, and midazolam for CYP3A4/5. This combination of probes has been validated in the Cooperstown 5+1 Cocktail (5+1).1 The use of the 5+1 cocktail provides information on the drug metabolizing enzymes that metabolize 90% of hepatically eliminated drugs for a fraction of the costs of the individual studies. Using a cocktail of biomarkers reduces the overall cost of drug interaction screening. The purpose of this study is to evaluate the effects of three Food and Drug Administration (FDA) approved oral antibiotics (azithromycin, telithromycin, and levofloxacin) on metabolism of other medications when taken together. This will be determined by the measuring the activity of drug metabolizing enzymes following administration of certain drug probes (caffeine, dextromethorphan, omeprazole, midazolam, and warfarin with vitamin K). A total of 16 subjects will complete four phases of the study: 1) Cooperstown 5+1 alone, 2) Azithromycin plus Cooperstown 5+1, 3) Telithromycin plus Cooperstown 5+1, and 4) Levofloxacin plus Cooperstown 5+1.

DETAILED DESCRIPTION:
Specific Aims

1. What is the purpose of this study? What question is it designed to answer?

   To compare the effect of azithromycin, telithromycin, and levofloxacin on activity of 7 hepatic drug metabolizing enzymes using the Cooperstown 5+1 Cocktail.

   Background
2. Why is this study important?

We have previously shown that a broad drug interaction screening can be performed using enzyme specific probes such as oral caffeine for CYP1A2, N-acetyltrasferase-2 (NAT-2), and xanthine oxidase (XO), warfarin plus vitamin K for CYP2C9, omeprazole for CYP 2C19, dextromethorphan for CYP2D6, and midazolam for CYP3A4/5. This combination of probes has been validated in the Cooperstown 5+1 Cocktail (5+1).1 The use of the 5+1 cocktail provides information on the drug metabolizing enzymes that metabolize 90% of hepatically eliminated drugs for a fraction of the costs of the individual studies. Using a cocktail of biomarkers reduces the overall cost of drug interaction screening. The FDA has indicated that the use of probe drugs can be done in place of specific drug interaction studies.2 This streamlines the detection of drug interactions and reduces costs. However, it is important to control for genetic polymorphism in drug interaction trials so that genetic makeup does not affect the outcome.

Experimental Design and Methods 3) Describe in detail the experimental design and methodology. What information will be collected and how will it be collected? Provide a description of the subject's participation from start to finish.

Prior to any procedure of the study each subject will provide written informed consent. All the subjects will be genotyped for CYP2D6, CYP2C9, and CYP2C19 after obtaining informed consent for pharmacogenomics. This is to distinguish poor metabolizers from extensive metabolizers.

Prestudy screening will be conducted within 4 weeks of the first study phase. Subjects will undergo a complete medical history, social history (including medication, alcohol, and tobacco use), physical examination, standard 12-lead electrocardiogram (ECG), and laboratory screening to assure that inclusion and exclusion criteria are met. The laboratory screening data to be obtained are: complete blood count, prothrombin time (PT), international normalized ratio (INR), macroscopic and microscopic urinalysis, electrolytes, blood urea nitrogen (BUN), serum creatinine, aspartate transaminase (AST), alanine transaminase (ALT), total bilirubin, and serum albumin. Women of childbearing potential (defined as premenopausal with no history of hysterectomy or tubal ligation) will undergo a serum pregnancy test during the screening visit and a urine pregnancy test prior to each phase of the study. Following enrollment, subjects will participate in each of the 4 study phases in a random order.

Study Design and Procedures This will be a randomized, crossover, open-label study. Prestudy screening will be conducted within 4 weeks of the first study phase. Screening visits will involve obtaining informed consent, medical history, social history, physical examination, ECG, and laboratory tests. Following enrollment, subjects will be randomized (and then crossed over) to 4 phases as described in Table 1.

Table 1. Study Design Study Drugs and Procedure Phase 1 (control) Cooperstown 5+1 Cocktail alone. The Cooperstown 5+1 Cocktail consists of the following components:

1. Caffeine (2 mg/kg orally, rounded to nearest 50 mg) with collection of a 12-hour urine.
2. Warfarin (10 mg + 10 mg vitamin K orally) with collection of plasma over 96 hours. Plasma collection times are at 0, 3, 6, 12, 24, 36, 48, 72 and 96 hours after dosing. The INR will be checked at 48 hours. If the INR is >1.7, 5 mg of vitamin K will be administered by mouth daily until the INR is 1.2.
3. Omeprazole (40 mg orally) with collection of a plasma sample 2 hours after dosing.
4. Dextromethorphan (30 mg orally) with collection of a 12-hour urine.
5. Midazolam (0.075 mg/kg orally) with collection of 8 plasma samples over 6 hours (only for Phase 1) to determine CYP3A activity (MDZ CL/F mL/min). Samples will be drawn immediately after midazolam administration (0 minute), then at 5 minute, 0.5, 1, 2, 4, 5 and 6 hours. Breathing, heart rate, and oxygen saturation will be monitored via pulse oximetry for the first 90 minutes after midazolam dose.

   Phase 2 Azithromycin 500 mg qAM for 3 days on an empty stomach. On day 4, the Cooperstown 5+1 Cocktail will be administered with a fourth dose of azithromycin given 2 hours after 5+1 administration.

   Phase 3 Telithromycin 800 mg qAM for 3 days on an empty stomach. On day 4, the Cooperstown 5+1 Cocktail will be administered with a fourth dose of telithromycin given 2 hours after 5+1 administration.

   Phase 4 Levofloxacin 750 mg qAM for 3 days on an empty stomach. On day 4, the Cooperstown 5+1 Cocktail will be administered with a fourth dose of levofloxacin given 2 hours after 5+1 administration.

   During the azithromycin, telithromycin, and levofloxacin phases, plasma samples for midazolam will be collected at 0.25, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, and 24 hours to allow for adequate sampling with drugs that potentially inhibit CYP3A. The 5+1 cocktail will be administered on day 4 after a minimum of 8-hour fasting.

   Subjects will not be allowed to eat until 2 hours after administration of study drugs (5+1 cocktail or antibiotic).

   Washout periods: One week after each phase except for the azithromycin phase is required to ensure the drug is completely eliminated from the body. Three weeks after the azithromycin phase is required since azithromycin has a longer half-life.

   Sample Collection and Analysis • For caffeine phenotyping, subjects will collect all of their urine for 12 hours after receiving the dose to determine CYP1A2 activity [(AFMU+1X+1U)/17U], NAT-2 [AFMU/(AFMU+1X+1U)], and XO [1U/(1X+1U)]. Urine will be acidified with ascorbic acid (in vitro) to prevent AFMU conversion.

   • For warfarin phenotyping, blood samples will be obtained at 0, 3, 6, 12, 24, 36, 48, 72 and 96 hours following warfarin plus vitamin K administration to determine CYP2C9 activity (S-warfarin CL/F, mL/min). For the first 12 hours, blood will be obtained through an intravenous (IV) catheter. Thereafter it will be via venipuncture.

   • For omeprazole phenotyping, one 15 mL blood sample will be drawn 2 hours after the oral omeprazole dose to determine CYP2C19 activity (OMP/5OH OMP).

   • For dextromethorphan phenotyping, subjects will collect all of their urine for 12 hours after receiving the dose to determine CYP2D6 activity (DM/DX).
   * For midazolam phenotyping, use of oral midazolam gives an assessment of inhibition of both gut and hepatic CYP3A.

     * For Phase 1 (5+1 cocktail alone), 8 blood samples (10 mL each) will be obtained immediately after midazolam administration (0 minute), then at 5 minutes, 0.5, 1, 2, 4, 5 and 6 hours to determine CYP3A activity (MDZ CL/F, mL/min).
     * During the azithromycin, telithromycin, and levofloxacin phases, blood samples will be collected at 0.25, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, and 24 hours (to allow for adequate sampling with drugs that potentially inhibit CYP3A).
   * All blood samples (except 15 mL for omeprazole) will be collected in duplicate in 10 mL EDTA-containing test tubes and centrifuged for 15 minutes at 2800 rpm.
   * Plasma and urine samples will be frozen at -80C until analysis.

   Data Analysis • Caffeine phenotyping assay: Urine aliquots will be assayed to determine urinary concentration of 1U, 1X, 17U, and AFMU. Urine aliquots will be analyzed at University of Missouri, Kansas City. Caffeine demethylation ratios will be used to express CYP1A2, NAT-2, and XO activity.

   • S- and R-warfarin phenotyping assay: S- and R-warfarin in plasma will be determined utilizing high performance liquid chromatography (HPLC) analysis at the University of North Carolina, Chapel Hill. Warfarin clearance will be determined using non-compartmental analysis. WinNonlin® 3.1 will be used for pharmacokinetic analyses.

   • Omeprazole phenotyping assay: Blood samples will be analyzed at the University of North Carolina, Chapel Hill, to determine plasma concentrations of OMP and 5OH OMP. The ratio of OMP and 5OH OMP at 2 hours following the oral dose of omeprazole will be used to describe CYP2C19 activity.

   • Dextromethorphan phenotyping assay: Urine aliquots will be analyzed at University of Missouri, Kansas City, to determine urinary concentrations of DM/DX. The dextromethorphan metabolic ratio will be used to describe CYP2D6 activity.

   • Midazolam phenotyping assay: Blood samples will be analyzed to determine plasma concentration of midazolam, 1-hydroxymidazolam, and 4-hydroxymidazolam. Analyses will be performed at Oneida Research Services, Inc. using a proprietary LC/MS/MS method. Midazolam clearance will be used to reflect CYP3A activity and clearance will be determined by using non-compartmental analysis of midazolam plasma concentration-time data. WinNonlin® 3.1 will be used for pharmacokinetic analyses.

   Statistical Analysis
   * Sample size: Using =0.05, four treatment phases, and =0.20 (power of 80%), an estimated sample size of sixteen volunteers will detect a 25% difference in metabolism.
   * Data will be analyzed using the FDA's standard bioequivalency testing.3 If the drug phases fall outside of the 0.8-1.25 range versus the control phase, BE will not be shown.

4) If the research is in part a treatment protocol, identify which parts are routine and which parts are being done solely for research.

This study is for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18 and 55 years.
* Ability to provide written informed consent.
* Willing to avoid all medications (other than the study drugs) which may inhibit or induce hepatic microsomal enzymes during the study period. This includes prescription and non-prescription medications, vitamins, herbal supplements, and nutriceuticals.
* Willing to avoid drinking more than the equivalence of one beer per day (one 12 ounce beer or equivalent alcohol intake) throughout the study period.
* Women of child-bearing potential who are willing to practice non-hormonal methods of contraception during all study phases.
* Willing to adhere to dietary restrictions as required during the study.

Exclusion Criteria:

* Clinically significant abnormal findings by history, physical exam, ECG, or laboratory testing.
* Elevated liver function tests twice above the upper limit of the normal range (males AST 0-50 U/L, ALT 0-60 U/L, GGT 11-50; females AST 0-40 U/L, ALT 0-50 U/L, GGT 7-32), or total bilirubin >1.3mg/dL.
* Baseline INR >1.2.
* Serum creatinine above the normal ranges
* Women who are pregnant, breastfeeding, and/or not using an acceptable form of non-hormonal contraception (barrier method or abstinence) during the study.
* History of gastrointestinal bleeding or peptic ulcer disease.
* Any condition that may affect drug absorption (e.g., gastrectomy, malabsorption syndromes).
* History of known hypersensitivity or serious adverse reaction to azithromycin, telithromycin, levofloxacin, midazolam, dextromethorphan, caffeine, omeprazole, heparin, warfarin, or vitamin K.
* Poor IV access as determined by an investigator.
* Current illicit drug use.
* History of tobacco use within 3 months of screening.
* Use of any drug known to inhibit or induce hepatic enzymes within 30 days of the first study phase.
* Regular alcohol intake exceeding 1 drink/day (1 drink = 5 ounces of wine or 12 ounces of beer or 1 ounce of hard liquor) within 1 months of screening.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study drug.
* Presence of any condition that the investigator feels would interfere with successful completion of the study.
* Poor metabolizers of CYP2D6, CYP2C9, and CYP2C19.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2004-11; Study Completion 2005-06

PRIMARY OUTCOMES:
Phenotype measures

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Bertino, Pharm.D., Principal Investigator — Bassett Healthcare